CLINICAL TRIAL: NCT04587557
Title: The Effects of Storytelling With or Without Social Contextual Information Regarding Eye Gaze and Visual Attention in Children With Autistic Spectrum Disorder and Typical Development: A Randomized, Controlled Eye-tracking Study
Brief Title: Storytelling With or Without Social Contextual Information in Children With Autistic Spectrum Disorder and Typical Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Kenneth N. K. Fong, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20160427001
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Autism Spectrum Disorder; Healthy
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ASD Group 1 - storytelling with social contextual information (Experimental): Storytelling with social contextual information for children with Autism Spectrum Disorder
  Interventions: Behavioral: Storytelling with social contextual information; Other: Children with ASD
- ASD Group 2 - storytelling without social contextual information (Active Comparator): Storytelling without social contextual information for children with Autism Spectrum Disorder
  Interventions: Behavioral: Storytelling without social contextual information; Other: Children with ASD
- TD Group 1 - storytelling with social contextual information (Experimental): Storytelling with social contextual information for typically developed children
  Interventions: Behavioral: Storytelling with social contextual information; Other: Children with TD
- TD Group 2 - storytelling without social contextual information (Active Comparator): Storytelling without social contextual information for typically developed children
  Interventions: Behavioral: Storytelling without social contextual information; Other: Children with TD

INTERVENTIONS:
Behavioral: Storytelling with social contextual information — Four out of 100 stories from a storytelling app (SAHK, 2013) that incorporated social contextual information, and inter-personal skills were selected. The intervention was in small group format, consisted of eight sessions across four weeks, two sessions per week, 30 minutes per session.
  Arms: ASD Group 1 - storytelling with social contextual information; TD Group 1 - storytelling with social contextual information
Behavioral: Storytelling without social contextual information — Four out of 100 stories from a storytelling app (SAHK, 2013) without social contextual information, and inter-personal skills were selected. The intervention was in small group format, consisted of eight sessions across four weeks, two sessions per week, 30 minutes per session.
  Arms: ASD Group 2 - storytelling without social contextual information; TD Group 2 - storytelling without social contextual information
Other: Children with ASD — Four out of 100 stories from a storytelling app (SAHK, 2013) were selected for children with ASD.
  Arms: ASD Group 1 - storytelling with social contextual information; ASD Group 2 - storytelling without social contextual information
Other: Children with TD — Four out of 100 stories from a storytelling app (SAHK, 2013) were selected for children with TD.
  Arms: TD Group 1 - storytelling with social contextual information; TD Group 2 - storytelling without social contextual information

SUMMARY:
This study was to examine the effects of storytelling with or without contextual information on children with autism spectrum disorder (ASD) and typical development (TD).

DETAILED DESCRIPTION:
This was a 2 x 2 x 2 randomized controlled trial with 52 children (26 with ASD and 26 with TD) recruited in the community and randomized into four groups: 1) ASD Group 1 - storytelling with contextual information; 2) ASD Group 2 - storytelling without contextual information; 3) TD Group 1 - storytelling with contextual information; 4) TD Group 2 - storytelling without contextual information. All stories were photo-based and static in nature. The only difference between Group 1 and Group 2 was that the stories included and did not include social contextual information, respectively. Training was delivered in small groups, with eight sessions across four weeks, two sessions per week, and 30 minutes per session. Participants' total fixation duration (TFD), total visit duration (TVD), and total fixation count (TFC) on human faces from 20 photos and a video were recorded using the Tobii eye tracker.

ELIGIBILITY:
Inclusion Criteria for children with ASD:

* 1) children aged between 6 and 12 years old;
* 2) had a previous diagnosis of ASD from medical professionals;
* 3) studied in mainstream primary school;
* 4) had a composite IQ score of 80 or above

Inclusion Criteria for children with TD:

* 1) children aged between 6 and 12 years old;
* 2) had no developmental disorder or intellectual disability;
* 3) attended primary school.

Exclusion Criteria:

* NA

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Eye gaze on the eye tracker | Change from baseline to 4 weeks
  Total fixation duration (TFD)
Eye gaze on the eye tracker | Change from baseline to 4 weeks
  Total visit duration (TVD)
Eye gaze on the eye tracker | Change from baseline to 4 weeks
  Total fixation count (TFC)

SECONDARY OUTCOMES:
Trail Making Test | Change from baseline to 4 weeks
  Trail Making Test A (TMT-A)
Trail Making Test | Change from baseline to 4 weeks
  Trail Making Test B (TMT-B)

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Department of Rehabilitation Sciences, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Upon request

REFERENCES:
- [Derived] Tang WYF, Fong KNK, Chung RCK. The Effects of Storytelling With or Without Social Contextual Information Regarding Eye Gaze and Visual Attention in Children with Autistic Spectrum Disorder and Typical Development: A Randomized, Controlled Eye-Tracking Study. J Autism Dev Disord. 2022 Mar;52(3):1257-1267. doi: 10.1007/s10803-021-05012-w. Epub 2021 Apr 28. PMID 33909213